CLINICAL TRIAL: NCT02260674
Title: A Phase 2a Randomized, Double-blind, Placebo-Controlled, Parallel-Group, Multi-center Study Investigating the Safety and Tolerability of JNJ-54861911 in Subjects With Early Alzheimer's Disease
Brief Title: A Safety and Tolerability Study of JNJ-54861911 in Participants With Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR105240; 54861911ALZ2002 (Other: Janssen Research & Development, LLC); 2014-002159-24 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; JNJ-54861911; Placebo
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Group 1 (Experimental): Participants will self-administer JNJ-54861911, two tablets of 5 milligram (mg) each for a total of 10 mg, orally, once daily, from Day 1 until Month 6.
  Interventions: Drug: JNJ-54861911, 10 milligram (mg)
- Treatment Group 2 (Experimental): Participants will self-administer JNJ-54861911, two tablets of 25 mg each for a total of 50 mg, orally, once daily, from Day 1 until Month 6.
  Interventions: Drug: JNJ-54861911, 50 mg
- Placebo (Placebo Comparator): Placebo matched to JNJ-54861911, orally, once daily, from Day 1 until Month 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54861911, 10 milligram (mg) — Participants will self-administer JNJ-54861911, two tablets of 5 mg each for a total of 10 mg, orally, once daily, from Day 1 until Month 6 in treatment group 1.
  Arms: Treatment Group 1
Drug: JNJ-54861911, 50 mg — Participants will self-administer JNJ-54861911, two tablets of 25 mg each for a total of 50 mg, orally, once daily, from Day 1 until Month 6 in treatment group 2.
  Arms: Treatment Group 2
Drug: Placebo — Placebo matched to JNJ-54861911, orally, once daily, from Day 1 until Month 6 in placebo group.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of JNJ-54861911 during 6 months of treatment in participants with early (predementia) alzheimer's disease (AD [degenerative disease of the brain characterized by the insidious onset of dementia, impairment of memory, judgment, attention span, and problem solving skills are followed by severe apraxias and a global loss of cognitive abilities]).

DETAILED DESCRIPTION:
This is a double-blind (neither the researchers nor the participants know what treatment the participant is receiving), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), randomized (study drug assigned by chance), multi-center (when more than one hospital or medical school team work on a medical research study), parallel-group study. The study consists of 3 Parts; Screening Phase of 90 days, double-blind Treatment Phase of 6 months and Follow-up Phase of 7 to 28 days following the last dose in Month 6. Eligible participants in the early (predementia) AD spectrum will be randomized to either Treatment group 1, 2 or placebo and participants who previously participated in study 54861911ALZ1005 will be enrolled in this study and will receive the same treatment as in study 54861911ALZ1005. The study duration for each participant will be approximately 10 months. Blood and cerebrospinal fluid (CSF) samples will be collected to evaluate the plasma pharmacokinetics of JNJ-54861911, as well as amyloid beta fragments. Participants' safety will be monitored throughout the study, including magnetic resonance imaging (MRI) and cognitive measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the early alzheimer's disease (AD) spectrum must have a global Clinical Dementia Rating Scale( CDR) score of 0 (asymptomatic at risk for AD) to 0.5 prodromal AD (pAD) inclusive
* Participants must have evidence of amyloid pathology by means of either: a) low Cerebrospinal Fluid (CSF) ABeta 1-42 levels at screening; b) a positive amyloid positron emission tomography (PET) scan at screening (depending on the site's PET capability) by visual read
* Participants must have a body mass index between 18 and 35 kilogram per square meter (kg/m^2), inclusive, at screening
* Participants must be otherwise healthy for their age group or medically stable with or without medication on the basis of physical examination, medical history, vital signs, and 12-lead ECG performed at screening or at baseline. If there are abnormalities, they must be consistent with the underlying illness in the study population and not a potential cause of cognitive impairment, with written concurrence with the sponsor's medical monitor
* Before randomization, a woman must be not of childbearing potential: postmenopausal (greater than or equal to [>=] 50 years of age with amenorrhea for at least 12 months; permanently sterilized [e.g., tubal occlusion, hysterectomy, bilateral salpingectomy]); or otherwise be incapable of pregnancy. In case of questionable status qualified personal of the sponsor should be consulted to decide on the potential for inclusion of the participant

Exclusion Criteria:

* Participant has evidence of any brain disease, other than potential very early signs of AD (e.g. mild hippocampal atrophy) or typical age-related changes (e.g. mild white matter hyperintensity on magnetic resonance imaging [MRI]) or any other abnormality (e.g. folic acid/Vitamin B12 deficiency) that could explain a possible cognitive deficit (including, but not limited to vascular encephalopathy or strokes including lacuna's (as imaged by cerebral MRI) and Major Depression (as defined by most current Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria)
* Participant has evidence of familial autosomal dominant AD. (Inclusion can be made upon written confirmation by sponsor, when the mutation is known and deemed not to be modulating Beta-secretase [BACE] cleavage)
* Participant with history or presence of significant depression as defined by the most current DSM criteria
* Participant has a clinically significant abnormal physical- or neurological examination, vital signs at screening or baseline (Day 1 predose)
* Participant has a history of or current liver or renal insufficiency; clinically significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, hematologic, rheumatologic, psychiatric, or metabolic disturbances (e.g. unstable situation needing monitoring or regular dose adaptations)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | up to 10 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Relationship Between Dose and Exposure of JNJ-54861911 With Safety | Month 1 up to Month 6
  Plasma and, if possible, CSF measurements will be taken to measure the concentration of JNJ-54861911. Population pharmacokinetic modeling (statistical modeling) will be used to derive individual pharmacokinetic parameters (e.g. Cmax, AUCtau, Tmax) in plasma and, if possible, in CSF. Incidence of adverse events and their timing of onset will be examined with regard to these concentrations to assess potential relationships between safety and exposure.
Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid Beta (ABeta) (1-37, 1-38, 1-40, 1-42) Levels and Soluble Amyloid Precursor Protein (sAPP) Fragments (sAPP-alpha, sAPP-beta), Total sAPP Levels | Baseline and Month 6
  The CSF samples will be obtained for measuring levels of different ABeta fragments such as ABeta 1-37, ABeta 1-38, ABeta 1-40, ABeta 1-42. ABeta fragments of different length are produced by cleavage of the APP by beta-secretase (BACE) and the gamma-secretase complex in the brain and excreted into CSF. For participants, who participated previously in study 54861911ALZ1005, the baseline CSF sample taken during that study may be used as baseline in this study.
Percent Change From Baseline in Plasma ABeta 1-40 Levels and sAPP Fragments (sAPP-alpha, sAPP-beta), Total sAPP Levels | Baseline and Month 6 (Day 168)
  Plasma samples will be obtained for measuring levels of different ABeta fragments such as ABeta 1-37, ABeta 1-38, ABeta 1-40, ABeta 1-42. ABeta fragments of different length are produced by cleavage of the APP by beta-secretase (BACE) and the gamma-secretase complex in the different peripheral tissues, including white blood cells and can be measured in Plasma.
Relationship Between Changes in CSF and Plasma ABeta Species and sAPP Fragments With Safety | Month 1 up to Month 6
  ABeta species and sAPP fragments in plasma and CSF will be measured. Incidence of adverse events and their timing of onset will be examined with regard to these concentrations to assess potential relationships between safety and changes in the ABeta species and sAPP fragments.
Maximum Plasma Concentration (Cmax) of JNJ-54861911 | Pre-dose on Day 1, post-dose on Day 28, 56, 84, 112, 140 and 168
  The Cmax is the maximum observed plasma concentration.
Time to Reach the Maximum Plasma or CSF concentration (Tmax) | Pre-dose on Day 1, post-dose on Day 28, 56, 84, 112, 140 and 168
  The Tmax is the time to reach the maximum plasma or CSF concentration.
Area Under the Plasma/CSF Concentration-time Curve From Time 0 to tau Hours Post Dosing (AUCtau) | Pre-dose on Day 1, post-dose on Day 28, 56, 84, 112, 140 and 168
  AUCtau is the area under the plasma/CSF concentration-time curve from time 0 to tau hours post dosing. Time tau is the dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (19):
- Belgium (2):
  - Ghent
  - Hoboken
- France (3):
  - Montpellier
  - Paris
  - Toulouse
- Germany (7):
  - Essen
  - Halle
  - Hamburg
  - Homburg
  - Lübeck
  - Tübingen
  - Ulm
- Amsterdam, Netherlands
- Spain (4):
  - Barcelona
  - Madrid
  - Terrasa Barcelona N/A
  - Valencia
- Sweden (2):
  - Mölndal
  - Stockholm

REFERENCES:
- [Derived] Novak G, Streffer JR, Timmers M, Henley D, Brashear HR, Bogert J, Russu A, Janssens L, Tesseur I, Tritsmans L, Van Nueten L, Engelborghs S. Long-term safety and tolerability of atabecestat (JNJ-54861911), an oral BACE1 inhibitor, in early Alzheimer's disease spectrum patients: a randomized, double-blind, placebo-controlled study and a two-period extension study. Alzheimers Res Ther. 2020 May 14;12(1):58. doi: 10.1186/s13195-020-00614-5. PMID 32410694